CLINICAL TRIAL: NCT04160572
Title: Sleep Schedule Intervention Study Among Night Shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wan-Ju Cheng, Physician, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMUH108-REC3-097
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Shift Work Schedule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning-evening sleep schedule (Experimental)
  Interventions: Behavioral: Morning sleep schedule; Behavioral: Evening sleep schedule
- Evening-morning sleep schedule (Active Comparator)
  Interventions: Behavioral: Morning sleep schedule; Behavioral: Evening sleep schedule

INTERVENTIONS:
Behavioral: Morning sleep schedule — sleep right after night shifts
Behavioral: Evening sleep schedule — sleep before night shifts

SUMMARY:
This study will recruit 60 night shift workers with shift work disorder. They will be invited to wear actigraphy for 3 weeks. In the first week the participants will sleep at the time they used to, and their chronotype will be determined by actigraphy and Munich Chronotype Questionnaire. In the second week the participants will be randomly assigned to morning sleep or evening sleep time, and will change to the other in the third week. We will compare sleepiness, sleep quality, daytime vigilance score changes using mixed method ANOVA. We will also examine the interaction effect of chronotype and sleep schedule on sleep-related outcome.

ELIGIBILITY:
Inclusion Criteria:

* Shift work disorder

Exclusion Criteria:

* Neuromuscular disorder
* Taking hypnotics
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Change from baseline score at the second and third week.
  Pittsburgh sleep quality index (PSQI), range from 0 (better) to 21 (worse)

SECONDARY OUTCOMES:
Daytime sleepiness | Change from baseline score at the start and end of each night shift.
  Karolinska Sleepiness Scale (KSS), range from 1 (better) to 9 (worse)
Alertness | Change from baseline score at the start and end of each night shift.
  Psychomotor vigilance test (PVT), reaction time (longer the worse) and lapses (larger the worse)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng WJ, Hang LW, Kubo T, Vanttola P, Huang SC. Impact of sleep timing on attention, sleepiness, and sleep quality among real-life night shift workers with shift work disorder: a cross-over clinical trial. Sleep. 2022 Apr 11;45(4):zsac034. doi: 10.1093/sleep/zsac034. PMID 35148396